CLINICAL TRIAL: NCT04967612
Title: Evaluation of Visual Perception Through Diffractive Optical Lens Designs by Virtual Implantation.
Brief Title: Visual Perception After Virtual Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PJV2002
Record Dates: First submitted 2021-07-07; First posted 2021-07-19 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual implantation of diffractive optical lens design A (Experimental)
  Interventions: Other: Virtual implantation
- Virtual implantation of diffractive optical lens design B (Experimental)
  Interventions: Other: Virtual implantation
- Virtual implantation of diffractive optical lens design C (Experimental)
  Interventions: Other: Virtual implantation

INTERVENTIONS:
Other: Virtual implantation — Temporary placement of virtual optical lens in the crystalline lens plane.

SUMMARY:
Evaluation of visual perception through diffractive optical lens designs by virtual implantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between and including 18 and 50 years of age;
* Healthy eyes;
* Dominant eye with a monocular CDVA ≥1.0 decimal (≤ 0.0 logMAR) without cycloplegia;
* Subject who has been informed of the consequences and constraints of the protocol and who has given his/her written informed consent;
* Negative COVID19 screening test prior to every trial visit.

Exclusion Criteria:

* Subjects of less than 18 or more than 50 years of age;
* Monocular CDVA of dominant eye < 1.0 decimal (> 0.0 logMAR) without cycloplegia;
* Subject unable to comply with the study protocol or likely to be non-cooperative during the study;
* Subject whose freedom is impaired by administrative or legal issues, or adult persons under legal protection or unable to give an informed consent;
* Pseudophakic subjects;
* Subjects, who are unable to fixate for a longer time, e.g. strabismus, nystagmus;
* Pathologic miosis;
* Intake of drugs affecting vision;
* Participation in another biomedical study in parallel, if it affects vision or if interactions with cycloplegia exist;
* Intolerance to or contraindication to cycloplegia, e.g. due to narrow angle of the anterior ocular chamber;
* Hyperopes with more than +6 D refraction.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Corrected distance visual acuity | during the intervention
  Evaluate visual acuity at distance following virtual implantation of diffractive optical lens designs

CONTACTS AND LOCATIONS:
Overall Officials: W Sickenberger, Prof, Principal Investigator — JenVis Research
Locations (1):
- JenVis Research, Jena, Germany